CLINICAL TRIAL: NCT03777631
Title: STroke Secondary Prevention With Catheter ABLation and EDoxaban for Patients With Non-valvular Atrial Fibrillation: STABLED Study
Acronym: STABLED
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nippon Medical School (Other)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Kazumi Kimura, Professor, Nippon Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LIX-DS-16018
Record Dates: First submitted 2018-11-03; First posted 2018-12-17 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Ischemic Stroke; Atrial Fibrillation Non-Rheumatic
Keywords: anticoagulation treatment; catheter ablation
MeSH Terms: conditions — Ischemic Stroke | interventions — Catheter Ablation

STUDY DESIGN:
Intervention Model Description: The included patients were randomly allocated to two groups: (1) Standard medical treatment group and (2) Catheter ablation additional group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard medical therapy group (No Intervention): The preferred anticoagulant is edoxaban. Antiarrhythmic drugs are administered as needed for the patient by well-trained cardiologists.
- Catheter ablation group (Active Comparator): Catheter ablation (CA) should be performed within 1-6 months from the onset of cerebral infarction. CA is based on pulmonary vein isolation, with atrial ablation as required. For conducting CA by a trained and experienced cardiologist, only institutions in which performed >100 CA annually were participated in the present study in principle.
  Interventions: Procedure: Catheter ablation

INTERVENTIONS:
Procedure: Catheter ablation — CA should be performed within 1-6 months from the onset of cerebral infarction. CA is based on pulmonary vein isolation, with atrial ablation as required.
  Arms: Catheter ablation group

SUMMARY:
Catheter ablation (CA) has been reported to reduce risk of stroke in patients with nonvalvular atrial fibrillation (NVAF) in retrospective studies, but risk and benefit of CA has not been well elucidated in NVAF with recent cerebral infarction in prospective randomized trials.

DETAILED DESCRIPTION:
In patients with NVAF, stroke is an independent risk factor for a subsequent cerebral infarction. Although anticoagulant therapy can effectively reduce thromboembolic events, the reported annual recurrence rate in NVAF and previous stroke patients in the "real-world" is not low even with appropriate antithrombotic treatment; 8.6% in patients with "guideline adherent" antithrombotic therapy and around 5% in patients treated with anticoagulant therapy. NVAF and recent stroke is high-risk population for stroke recurrence even with anticoagulant therapy, and developing optimal secondary prevention strategy is an urgent task.

Catheter ablation (CA) is now widely used to treat symptoms related to NVAF. Some retrospective studies showed a beneficial effect of CA for stroke prevention using age-/sex-matching or propensity-score matching. Moreover, CA have a potential to improve survival or prevent heart failure development in patients with AF. However, the effect of CA for secondary stroke prevention or impact of CA for NVAF patients with recent ischemic stroke for survival or developing heart failure has not been evaluated in a prospective randomized trial. Therefore, in the present study, we intend to compare two groups of patients with NVAF with a history of cerebral infarction: a group receiving standard medical therapy (control group) and a group receiving standard medical therapy plus CA (CA group).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥20 or ≤85 years at time of giving informed consent
* Nonvalvular atrial fibrillation
* History of stroke in previous 6 months
* Current or planned treatment with edoxaban
* Modified Rankin scale ≤3

Exclusion Criteria:

* Symptomatic paroxysmal AF resistant to anti-arrhythmic drugs
* Presence of left atrial thrombus and left atrial appendage on transthoracic echocardiography, computed tomography or magnetic resonance imaging
* Unable to take anticoagulation therapy for any reason, including tendency to bleed or considered at high risk for bleeding from anticoagulation therapy.
* Presence of severe renal disorder (estimated creatinine clearance <30 mL/min by Cockroft-Gault equation)
* Previous CA or surgical intervention for AF
* History of treatment with a left atrial appendage closure device
* Left atrial diameter ≥55 mm on transthoracic echocardiography
* Ejection fraction ≤35% on transthoracic echocardiography
* Persistent AF for ≥10 years
* Pregnant or possibility of pregnancy
* Unlikely to complete the study, such as due to progressive malignant tumor
* Participating or planning to participate in another clinical trial
* Unwilling to participates
* Judged as incompatible for the study by the investigators

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Composite of recurrence of cerebral infarction, systemic embolism, all-cause death, hospitalization for heart failure. | Up to 6 years
  Composite of recurrence of cerebral infarction, systemic embolism, all-cause death, hospitalization for heart failure.

SECONDARY OUTCOMES:
Recurrence of cerebral infarction | Up to 6 years
  Recurrence of cerebral infarction
Systemic embolism | Up to 6 years
  Symptomatic systemic embolism to other regions than brain, e.g. peripheral or visceral arteries
All-cause death | Up to 6 years
  All-cause death
Cardiovascular death | Up to 6 years
  Cardiovascular death
Hospitalization for heart failure | Up to 6 years
  Hospitalization for heart failure
Any bleeding | Up to 6 years
  Any bleeding
Intracranial hemorrhage | Up to 6 years
  Intracranial hemorrhage
Composite events | Up to 6 years
  all-cause death, onset of stroke, systemic embolism, hospitalization for heart failure, and serious adverse event caused by CA
The rate of and related factors to discontinuation of Edoxaban | Up to 6 years
  The rate of and related factors to discontinuation of Edoxaban
Recurrence of cerebral infarction in patients with or without discontinuation of Edoxaban | Up to 6 years
  Recurrence of cerebral infarction in patients with or without discontinuation of Edoxaban

OTHER OUTCOMES:
Incidence of treatment-emergent adverse events (safety and tolerability) | Within 1 month after CA
  Incidence of treatment-emergent adverse events (safety and tolerability)
Incidence of all adverse events, not restricted to CA maneuver-related adverse events | Within 1 month after CA
  Incidence of all adverse events, not restricted to CA maneuver-related adverse events
Drug reaction to edoxaban | Up to 6 years
  Drug reaction to edoxaban

CONTACTS AND LOCATIONS:
Overall Officials: Kazumi Kimura, M.D., Ph.D, Principal Investigator — Department of Neurology, Nippon Medical School
Locations (46):
- Japan (46):
  - Ichinomiyanishi Hospital, Aichi
  - Hirosaki Stroke and Rehabilitation Center, Aomori
  - Hirosaki University Hospital, Aomori
  - Kimitsu Chuo Hospital, Chiba
  - New Tokyo Heart Clinic, Chiba
  - New Tokyo Hospital, Chiba
  - Nippon Medical School Chiba Hokusoh Hospital, Chiba
  - Kokura Memorial Hospital, Fukuoka
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Ogaki Municipal Hospital, Gifu
  - Brain Attack Center Ota Memorial Hospital, Hiroshima
  - Fukuyama Cardiovascular Hospital, Hiroshima
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Hiroshima University Hospital, Hiroshima
  - Suiseikai Kajikawa Hospital, Hiroshima
  - Teine Keijinkai Hospital, Hokkaido
  - Hyogo Brain and Heart Center, Hyōgo
  - Hyogo College of Medicine College Hospital, Hyōgo
  - Kitaharima medical center, Hyōgo
  - Odawara Cardiovascular Hospital, Kanagawa
  - Seisho Hospital, Kanagawa
  - National Hospital Organization Kanazawa Medical Center, Kanazawa
  - Kumamoto Red Cross Hospital, Kumamoto
  - Saiseikai Kumamoto Hospital, Kumamoto
  - Iwate Medical University, Morioka
  - Iwate Prefectural Central Hospital, Morioka
  - Nagasaki University Hospital, Nagasaki
  - Tenri Hospital, Nara
  - Okayama Red Cross Hospital, Okayama
  - National Cerebral and Cardiovascular Center, Osaka
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka General Medical Center, Osaka
  - Saga Medical Center Koseikan, Saga
  - Saitama Medical Center, Saitama
  - Saitama Medical University International Medical Center, Saitama
  - Dokkyo Medical University Hospital, Tochigi
  - Jichi Medical University Hospital, Tochigi
  - Jikei University Hospital, Tokyo
  - Juntendo University Hospital, Tokyo
  - Kyorin University Hospital, Tokyo
  - Nippon Medical School, Tokyo
  - NTT Medical Center Tokyo, Tokyo
  - Showa University Koto Toyosu Hospital, Tokyo
  - Tokyo Women's Medical University Hospital, Tokyo
  - Tsuruoka Kyoritsu Hospital, Yamagata
  - Tsuruoka Municipal Shonai Hospital, Yamagata

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sakamoto Y, Nishiyama Y, Iwasaki YK, Daida H, Toyoda K, Kitagawa K, Okumura K, Kusano K, Hagiwara N, Fujimoto S, Miyamoto S, Otsuka T, Iguchi Y, Kanamaru T, Yamamoto T, Kaburagi J, Kimura T, Matsumoto T, Kimura K, Shimizu W; STABLED Study Investigators. Design and rationale of the STroke secondary prevention with catheter ABLation and EDoxaban clinical trial in patients with non-valvular atrial fibrillation: The STABLED study. J Cardiol. 2019 Dec;74(6):539-542. doi: 10.1016/j.jjcc.2019.06.002. Epub 2019 Jul 20. PMID 31337525